CLINICAL TRIAL: NCT03028545
Title: Representations, Strategies and Identity Redefinition in the Recovery Process: Exploratory Study
Brief Title: Representations and Strategies for Recovery
Acronym: EPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A01049-42
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Schizophrenia, Undifferentiated; Anorexia; Bipolar Disorders; Personality Disorders
Keywords: schizophrenia; anorexia; bipolar disorders; personality disorders
MeSH Terms: conditions — Schizophrenia; Disorders of Sex Development; Anorexia; Bipolar Disorder; Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- schizophrenia (Other): Exploring and understanding, through a multidisciplinary exploration (medical, anthropological and sociological) representations and recovery strategies in schizophrenia
  Interventions: Behavioral: Collection of the individual narrative, semi-directed interviews
- bipolar disorders (Other): Exploring and understanding, through a multidisciplinary exploration (medical, anthropological and sociological) representations and recovery strategies in bipolar disorders
  Interventions: Behavioral: Collection of the individual narrative, semi-directed interviews
- eating disorders (Other): Exploring and understanding, through a multidisciplinary exploration (medical, anthropological and sociological) representations and recovery strategies in eating disorders
  Interventions: Behavioral: Collection of the individual narrative, semi-directed interviews
- personality disorders (Other): Exploring and understanding, through a multidisciplinary exploration (medical, anthropological and sociological) representations and recovery strategies in personality disorders
  Interventions: Behavioral: Collection of the individual narrative, semi-directed interviews

INTERVENTIONS:
Behavioral: Collection of the individual narrative, semi-directed interviews — Visit one : individual interview Individual narrative Passing Psychometric Measurement Scales of Recovery: Score at Warwick and Wellness Scale Andreasen scale score Visit two Focus group

SUMMARY:
In the recent context of deinstitutionalization and longitudinal studies pointing to a large number of positive long-term outcommes for people affected by a psychiatric disorder (schizophrenia, bipolar disorder, eating disorder, severe personality disorder, etc.), the possibility of overcoming the consequences of a psychiatric pathology emerges as a solid fact. Therefore, the existence of this possibility calls for the identification of the determinants underlying of the various outcomes over time of those affected by a severe psychiatric disorder, in particular those likely to underpin the most positive developments.

While it is well known from a medical point of view that certain dimensions affect the prognosis of persons affected by a severe psychiatric disorder (such as the persistence of negative symptoms or cognitive disorders in schizophrenic disorders), prognosis from a purely medical perspective (and putting aside the role of the person and his environment) seems to be able to account only for a modest proportion of the prognosis of people affected by a serious psychiatric disorder.

It is this fact that has gradually led to the emergence of complementary models capable of enriching the understanding of the determinants of the future of people affected by a severe psychiatric disorder, in particular models inviting to separate "becoming of the person" from the " psychiatric disorder "to take into account the" personal role of the person "in his or her own healing. This perspective is the "recovery" perspective.

Recovery process is defined as a personal trajectory which includes the person's experiences and the reactions of his / her environment following the installation of a psychiatric disorder, which can support a mode of release of the status of "psychiatric patient". Recovery thus implies an "approach underpinned by the understanding of the human response to pathology" (Noiseux) and, one might add, of its environment.

However, while these studies point to a number of crucial dimensions involved in the recovery of a severe psychiatric disorder, one of the important limitations of these studies is the distance from any psychopathological consideration, thus setting aside the possibility of specific processes of recovery depending of the pathology. The identification of recurrent experiential logics specific to the various psychiatric disorders therefore appears to be an important field of investigation. It would potentially be able to guide the development of new therapeutic devices based on the recovery model.

DETAILED DESCRIPTION:
1. Elaboration of a semi directed grid (exploratory phase)
2. Collection of individual narratives
3. Data analysis, according to IPA method (interpretative phenomenological analysis)

   * On the basis of individual narratives
   * On the basis of a focus group
4. Publication of results

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Psychiatric diagnosis according to DSM V critera of schizophrenia, eating disorder, bipolar disorder, personality disorder
* In recovery scale
* Informed of their diagnosis

Exclusion Criteria:

* Acute psychiatric state
* Poor understanding of french language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Collection of individual narratives to understand the recovery process | one year
  Semi-directed maintenance grid

SECONDARY OUTCOMES:
Change from baseline in the Quality of Well-Being at one year | one year
  Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS)
Change from baseline in measures of psychological recovery at one year | one year
  Stages of recovery instrument (STORI ANDREASEN)

CONTACTS AND LOCATIONS:
Overall Officials: MARTIN BRICE, MD/PhD, Principal Investigator — CH LE VINATIER
Locations (1):
- Vial Veronique, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No